CLINICAL TRIAL: NCT06892522
Title: A Phase 1/2, Open-Label, Platform Study to Evaluate Safety and Efficacy of Etentamig Monotherapy or Etentamig Combinations in Subjects With Multiple Myeloma
Brief Title: A Study to Assess Change in Disease Activity and Adverse Events (AE)s in Adult Participants With Multiple Myeloma Receiving Etentamig (ABBV-383) as an Intravenous (IV) Infusion Alone or in Combination With Oral, IV, Subcutaneous Daratumumab; Lenalidomide; Dexamethasone; Carfilzomib
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-059; 2024-515770-27-00 (Other: EU CT)
Record Dates: First submitted 2025-03-19; First posted 2025-03-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma, Etentamig, ABBV-383, Cancer; Daratumumab; Lenalidomide; Dexamethasone; Carfilzomib
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Lenalidomide; Dexamethasone; daratumumab; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Substudy 1: Etentamig Dose Escalation (Experimental): Participants will receive escalating etentamig in combination with daratumumab, and lenalidomide (DR), as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Lenalidomide; Drug: Daratumumab
- Substudy 1: Etentamig Dose Expansion Dose Level 1 (Experimental): Participants will receive dose level 1 of etentamig in combination with DR, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Lenalidomide; Drug: Daratumumab
- Substudy 1: Etentamig Dose Expansion Dose Level 2 (Experimental): Participants will receive dose level 2 of etentamig in combination with DR, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Lenalidomide; Drug: Daratumumab
- Substudy 1: Comparator (Experimental): Participants will receive daratumumab, lenalidomide, and dexamethasone (DRd), as part of the approximately 130 month study duration.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Daratumumab
- Substudy 2: Etentamig Dose Escalation (Experimental): Participants will receive escalating etentamig, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig
- Substudy 2: Etentamig Dose Expansion Dose Level 1 (Experimental): Participants will receive dose level 1 of etentamig, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig
- Substudy 2: Etentamig Dose Expansion Dose Level 2 (Experimental): Participants will receive dose level 2 of etentamig, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig
- Substudy 2: Comparator (Experimental): Participants will receive lenalidomide (R), as part of the approximately 130 month study duration.
  Interventions: Drug: Lenalidomide
- Substudy 3: Etentamig Dose Escalation (Experimental): Participants will receive escalating etentamig in combination with carfilzomib, and dexamethasone (Kd), as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Dexamethasone; Drug: Carfilzomib
- Substudy 3: Etentamig Dose Expansion Dose Level 1 (Experimental): Participants will receive dose level 1 of etentamig in combination with Kd, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Dexamethasone; Drug: Carfilzomib
- Substudy 3: Etentamig Dose Expansion Dose Level 2 (Experimental): Participants will receive dose level 2 of etentamig in combination with Kd, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Dexamethasone; Drug: Carfilzomib
- Substudy 3: Comparator (Experimental): Participants will receive daratumumab, carfilzomib, and dexamethasone (DKd), as part of the approximately 130 month study duration.
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Carfilzomib
- Substudy 4: Etentamig Dose Escalation (Experimental): Participants will receive escalating etentamig in combination with R, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Lenalidomide
- Substudy 4: Etentamig Dose Expansion Dose Level 1 (Experimental): Participants will receive dose level 1 of etentamig in combination with R, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Lenalidomide
- Substudy 4: Etentamig Dose Expansion Dose Level 2 (Experimental): Participants will receive dose level 2 of etentamig in combination with R, as part of the approximately 130 month study duration.
  Interventions: Drug: Etentamig; Drug: Lenalidomide

INTERVENTIONS:
Drug: Etentamig — Intravenous (IV) Infusion
  Arms: Substudy 1: Etentamig Dose Escalation; Substudy 1: Etentamig Dose Expansion Dose Level 1; Substudy 1: Etentamig Dose Expansion Dose Level 2; Substudy 2: Etentamig Dose Escalation; Substudy 2: Etentamig Dose Expansion Dose Level 1; Substudy 2: Etentamig Dose Expansion Dose Level 2; Substudy 3: Etentamig Dose Escalation; Substudy 3: Etentamig Dose Expansion Dose Level 1; Substudy 3: Etentamig Dose Expansion Dose Level 2; Substudy 4: Etentamig Dose Escalation; Substudy 4: Etentamig Dose Expansion Dose Level 1; Substudy 4: Etentamig Dose Expansion Dose Level 2
Drug: Lenalidomide — Oral Capsule
  Arms: Substudy 1: Comparator; Substudy 1: Etentamig Dose Escalation; Substudy 1: Etentamig Dose Expansion Dose Level 1; Substudy 1: Etentamig Dose Expansion Dose Level 2; Substudy 2: Comparator; Substudy 4: Etentamig Dose Escalation; Substudy 4: Etentamig Dose Expansion Dose Level 1; Substudy 4: Etentamig Dose Expansion Dose Level 2
Drug: Dexamethasone — IV Injection
  Arms: Substudy 1: Comparator; Substudy 3: Comparator; Substudy 3: Etentamig Dose Escalation; Substudy 3: Etentamig Dose Expansion Dose Level 1; Substudy 3: Etentamig Dose Expansion Dose Level 2
Drug: Daratumumab — Subcutaneous Injection
  Arms: Substudy 1: Comparator; Substudy 1: Etentamig Dose Escalation; Substudy 1: Etentamig Dose Expansion Dose Level 1; Substudy 1: Etentamig Dose Expansion Dose Level 2; Substudy 3: Comparator
Drug: Dexamethasone — Oral Tablet
  Arms: Substudy 1: Comparator; Substudy 3: Comparator; Substudy 3: Etentamig Dose Escalation; Substudy 3: Etentamig Dose Expansion Dose Level 1; Substudy 3: Etentamig Dose Expansion Dose Level 2
Drug: Carfilzomib — IV Infusion
  Arms: Substudy 3: Comparator; Substudy 3: Etentamig Dose Escalation; Substudy 3: Etentamig Dose Expansion Dose Level 1; Substudy 3: Etentamig Dose Expansion Dose Level 2

SUMMARY:
Multiple myeloma (MM) is a cancer of the blood's plasma cells. The cancer is typically found in the bones and bone marrow (the spongy tissue inside of the bones) and can cause bone pain, fractures, infections, weaker bones, and kidney failure. Treatments are available, but MM can come back (relapsed) or may not get better (refractory) with treatment. This is a study to determine the safety, efficacy, and pharmacokinetics of Etentamig in adult participants with MM.

Etentamig is an investigational drug being developed for the treatment of MM. This study is broken into 4 substudies and each substudy consists of a dose escalation phase and dose expansion phase. Participants will receive escalating doses of etentamig alone or in combination with daratumumab and lenalidomide (DR), carfilzomib and dexamethasone (Kd) or lenalidomide (R). This will be followed by etentamig at the dose levels established during the escalation phases alone or in combination with DR, Kd, R. The participants can also receive daratumumab, lenalidomide and dexamethasone (DRd), R, or daratumumab, carfilzomib, and dexamethasone (DKd) as a comparator in the dose expansion phases. Around 440 adult participants with MM will be enrolled at approximately 50 sites worldwide

In all substudies, participants will receive escalating doses of etentamig as Intravenous (IV) infusions, alone or in combination with DR, R or Kd, followed by IV infusions of etentamig at the dose levels established during the escalation phases alone or in combination with IV and oral DRd, DKd, or R. The study duration is approximately 130 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eastern cooperative oncology group (ECOG) performance of <= 1.
* Confirmed diagnosis of multiple myeloma (MM) according to the International Myeloma Working Group (IMWG) diagnostic criteria with either newly diagnosed or relapsed or refractory (RR) MM, depending on the substudy.

Exclusion Criteria:

* Participant who has known active central nervous system involvement of MM.
* Participant who has known active infection as outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2036-02 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE)s | Up to Approximately 130 Months
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Substudy 1: Dose-Limiting Toxicity (DLT) of Etentamig + Daratumumab and Lenalidomide (DR) in Participants with Transplant-Ineligible Newly Diagnosed Multiple Myeloma (TI NDMM) | Up to Approximately 8 weeks
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Substudy 2: DLT of Etentamig Monotherapy as Maintenance in Participants with Transplant-Eligible Newly Diagnosed Multiple Myeloma (TE NDMM) | Up to Approximately 8 Weeks
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Substudy 3: DLT of Etentamig +Carfilzomib and Dexamethasone (Kd) Combination in Participants with Relapsed or Refractory Multiple Myeloma (RR MM) | Up to Approximately 8 Weeks
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Substudy 4: DLT of Etentamig plus Lenalidomide when Given as Maintenance in Participants with TE NDMM | Up to Approximately 8 Weeks
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.

SECONDARY OUTCOMES:
Substudy 1, 2, 3, 4: Complete Response Rate | Up to Approximately 1 Year
  Complete response rate is defined as complete response (CR), stringent complete response (sCR) as assessed by the international myeloma working group (IMWG) 2016 criteria for MM.
Substudy 1, 2, 3, 4: Overall Response Rate (ORR) | Up to Approximately 1 Year
  The ORR is defined as the percentage of participants who achieve a best overall response of confirmed PR or better determined by IMWG criteria, prior to the initiation of subsequent myeloma therapy.
Substudy 1, 2, 3, 4: Progression Free Survival (PFS) | Up to Approximately 130 Months
  PFS is defined as the number of days from the date of first dose to the date of earliest disease progression (determined by the IMWG) or death.
Substudy 1, 2, 3, 4: Duration of Response (DOR) | Up to Approximately 130 Months
  DOR is defined as the time from the date of first response to the earliest occurrence of progressive disease, or death, whatever occurs first.
Substudy 1, 2, 3, 4: Time-to-Progression (TTP) | Up to Approximately 130 Months
  TTP will be defined as the number of days from the date of first dose to the date of earliest disease progression.
Substudy 1, 2, 3, 4: Minimal Residual Disease (MRD) negativity | Up to Approximately 52 Weeks
  The MRD negativity rate is defined as the proportion of participants who achieve MRD negative status.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (24):
- United States (7):
  - Colorado Blood Cancer Institute /ID# 273129, Denver, Colorado
  - Winship Cancer Institute of Emory University /ID# 274830, Atlanta, Georgia
  - Weill Cornell Medical College /ID# 272517, New York, New York
  - University of North Carolina at Chapel Hill /ID# 274667, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute /ID# 276193, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 274847, Winston-Salem, North Carolina
  - Oncology Hematology Care - Kenwood /ID# 272918, Cincinnati, Ohio
- Australia (8):
  - Coffs Harbour Health Campus /ID# 272010, Coffs Harbour, New South Wales
  - Port Macquarie Base Hospital /ID# 275925, Port Macquarie, New South Wales
  - Westmead Hospital /ID# 271880, Westmead, New South Wales
  - Icon Cancer Care - South Brisbane /ID# 271836, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 272629, Adelaide, South Australia
  - St Vincent's Hospital - Melbourne /ID# 276451, Fitzroy, Victoria
  - Peter MacCallum Cancer Centre /ID# 272024, Melbourne, Victoria
  - The Perth Blood Institute - West Perth /ID# 272469, West Perth, Western Australia
- Israel (5):
  - Soroka Medical Center /ID# 271367, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 271366, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus- Haifa /ID# 271364, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 271362, Jerusalem
  - Rabin Medical Center. /ID# 271365, Petah Tikva
- Japan (3):
  - Nagoya City University Hospital /ID# 273529, Nagoya, Aichi-ken
  - University Hospital Kyoto Prefectural University of Medicine /ID# 275713, Kyoto, Kyoto
  - The University of Osaka Hospital /ID# 275791, Suita-shi, Osaka
- Hammersmith Hospital /ID# 274615, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-059